CLINICAL TRIAL: NCT03639493
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerabillity of CJ-30060 in Healthy Male Subjects
Brief Title: Bioequivalence Study of CJ-30060 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_EXR_103
Record Dates: First submitted 2018-08-09; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Amlodipine, Valsartan Drug Combination; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: receive Exforge® tab 10/160mg, Crestor® tab 20mg
  * Period 2: receive CJ-30060 10/160/20mg
  Interventions: Drug: Exforge® tab 10/160mg, Crestor® tab 20mg; Drug: CJ-30060 10/160/20mg
- Sequence 2 (Experimental): * Period 1: receive CJ-30060 10/160/20mg
  * Period 2: receive Exforge® tab 10/160mg, Crestor® tab 20mg
  Interventions: Drug: Exforge® tab 10/160mg, Crestor® tab 20mg; Drug: CJ-30060 10/160/20mg

INTERVENTIONS:
Drug: Exforge® tab 10/160mg, Crestor® tab 20mg — Co-administration of Amlodipine 10mg/ Valsartan 160mg(combination drug) and Rosuvastatin 20mg
Drug: CJ-30060 10/160/20mg — Fixed-dose combination drug containing Amlodipine 10mg and Valsartan 160mg and Rosuvastatin 20mg

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 10/160mg, Crestor® 20mg in healthy male volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 10/160mg, Crestor® 20mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 20 to 45 years at screening
* BMI: 18 ~ 29.9kg/m^2
* Body weight ≥ 50kg
* Subjects who decided to participate in the study and signed informed consent form voluntarily after receiving detailed explanation of the study and fully understanding

Exclusion Criteria:

* Subjects who had a medical history of severe cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrinological, immunological, dermatological or neuropsychological disease
* Subjects who have symptoms of an acute disease within 28 days before first administration
* Subjects who have clinically significant active, chronic disease
* Subjects who fall under the criteria below in laboratory test

  * AST/ALT > UNL (upper normal limit) x 2
  * Total bilirubin > UNL x 1.5
  * CrCL < 50mL/min
  * CPK > UNL x 2.5
* Subjects with clinically significant low blood pressure at screening test (systolic blood pressure is less than 100 mmHg or diastolic blood pressure is less than 60 mmHg)
* Subjects with any positive reaction in HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL tests

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Cmax of amlodipine | Up to 144 hours post-dose
Cmax of valsartan | Up to 144 hours post-dose
Cmax of rosuvastatin | Up to 144 hours post-dose
AUClast of amlodipine | Up to 144 hours post-dose
AUClast of valsartan | Up to 144 hours post-dose
AUClast of rosuvastatin | Up to 144 hours post-dose

SECONDARY OUTCOMES:
AUCinf of amlodipine, valsaran, rosuvastatin | Up to 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No